CLINICAL TRIAL: NCT05847933
Title: A Pilot Study on the Influence of Temporo-occipital Transcranial Magnetic Brain Stimulation on Aversive Episodic Memory Performance
Brief Title: Influence of Temporo-occipital Transcranial Magnetic Brain Stimulation on Aversive Episodic Memory Performance
Acronym: SAME
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prof. Dominique de Quervain, MD (Other)
Responsible Party: Sponsor-Investigator, Prof. Dominique de Quervain, MD, Director Division of Cognitive Neuroscience, University of Basel
Organization: University of Basel (Other)
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: 2023-00392
Record Dates: First submitted 2023-04-14; First posted 2023-05-08 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Memory, Episodic
Keywords: memory; Transcranial magnetic brain stimulation; emotional valence
MeSH Terms: conditions — Recurrence | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (10):
- cTBS 50 Hz experiment (Experimental): Active brain stimulation on the temporo-occipital cortex using the cTBS 50 Hz protocol.
  Interventions: Device: rTMS (cTBS 50Hz experiment)
- cTBS sham (Sham Comparator): Sham brain stimulation on the temporo-occipital cortex using the cTBS 50Hz protocol pattern
  Interventions: Device: rTMS (cTBS sham)
- cTBS 50Hz active control (Active Comparator): Active brain stimulation on the right superior frontal cortex using the cTBS 50 Hz protocol
  Interventions: Device: rTMS (cTBS 50 Hz active control)
- High frequency (Experimental): Active brain stimulation on the temporo-occipital cortex using the 20Hz protocol
  Interventions: Device: rTMS (high frequency)
- Low frequency (Experimental): Active brain stimulation on the temporo-occipital cortex using the 1Hz protocol
  Interventions: Device: rTMS (low frequency)
- cTBS 30Hz (Experimental): Active brain stimulation on the temporo-occipital cortex using the cTBS 30 Hz protocol.
  Interventions: Device: rTMS (cTBS 30 Hz)
- cTBS 30 Hz Active control (Active Comparator): Active brain stimulation on the right superior frontal cortex using the cTBS 30 Hz protocol
  Interventions: Device: rTMS ( cTBS 30 Hz active control)
- High frequency Active control (Active Comparator): Active brain stimulation on the right superior frontal cortex using the 20 Hz online protocol
  Interventions: Device: rTMS (high frequency active control)
- Low frequency Active control (Active Comparator): Active brain stimulation on the right superior frontal cortex using the 1 Hz offline protocol
  Interventions: Device: rTMS (low frequency active control )
- High frequency sham (Sham Comparator): Brain stimulation on the dominant temporo-occipital cortex using 10% maximum system output (MSO) and 20 Hz online protocol.
  Interventions: Device: rTMS (high frequency sham)

INTERVENTIONS:
Device: rTMS (cTBS 50Hz experiment) — rTMS using cTBS protocol with the following characteristics:
  * Frequency: trains of 50 Hz (3 pulses) every 200ms (frequency of 5 Hz, in the range of theta band)
  * Intensity: 80% of resting motor threshold (rMT)
  * Location: consecutively on the left and right temporo-occipital cortex (MNI coordinates: left hemisphere: -50, -72, 4; right hemisphere:50, -66, 0)
  * Duration: 40 seconds for each hemisphere, 80 seconds in total.
  * Timing: Immediately before viewing pictures in pictorial memory task (off-line)
  Arms: cTBS 50 Hz experiment
Device: rTMS (cTBS sham) — rTMS using cTBS protocol with the following characteristics:
  * Frequency: trains of 50 Hz (3 pulses) every 200ms (frequency of 5 Hz, in the range of theta band)
  * Intensity: 0%
  * Location: consecutively on the left and right temporo-occipital cortex (MNI coordinates: left hemisphere: -50, -72, 4; right hemisphere:50, -66, 0)
  * Duration: 40 seconds for each hemisphere, 80 seconds in total.
  * Timing: Immediately before viewing pictures in pictorial memory task (off-line)
  Arms: cTBS sham
Device: rTMS (cTBS 50 Hz active control) — rTMS using cTBS protocol with the following characteristics:
  * Frequency: trains of 50 Hz (3 pulses) every 200ms (frequency of 5 Hz, in the range of theta band)
  * Intensity: 80% of resting motor threshold (rMT)
  * Location: Right superior frontal cortex
  * Duration: 40 seconds for each hemisphere, 80 seconds in total.
  * Timing: Immediately before viewing pictures in pictorial memory task (off-line)
  Arms: cTBS 50Hz active control
Device: rTMS (high frequency) — rTMS using high frequency protocol with the following characteristics:
  * Frequency: 20 Hz
  * Intensity: 120% of rMT for rMT < 54% & 65% of MSO for rMT ≥ 54%
  * Location: temporo-occipital cortex of the dominant brain hemisphere
  * Duration: 20 minutes, continuously
  * Timing: During the pictorial memory task (on-line) 1 second stimulation and 14 seconds inter-train interval for 76 trains resulting in a total of 1520 pulses.
  Arms: High frequency
Device: rTMS (low frequency) — rTMS using Low frequency protocol with the following characteristics:
  * Frequency: 1 Hz
  * Intensity: 110% of rMT
  * Location: temporo-occipital cortex of dominant brain hemisphere (MNI left hemisphere: -50, -72, 4; right hemisphere:50, -66, 0)
  * Duration: 30 minutes, continuously
  * Timing: Starting 10 minutes before and continuing during the picture viewing and valence rating of the pictures of the memory task (on-line).
  Arms: Low frequency
Device: rTMS (high frequency sham) — * Frequency: 20 Hz
  * Intensity: 10% of MSO
  * Location: temporo-occipital cortex of the dominant brain hemisphere
  * Duration: 20 minutes, continuously
  * Timing: During the pictorial memory task (on-line) 1 second stimulation and 14 seconds inter-train interval for 76 trains resulting in a total of 1520 pulses.
  Arms: High frequency sham
Device: rTMS (high frequency active control) — * Frequency: 20 Hz
  * Intensity: 120% of rMT for rMT < 54% & 65% of MSO for rMT ≥ 54%
  * Location: right superior frontal cortex of the dominant brain hemisphere
  * Duration: 20 minutes, continuously
  * Timing: During the pictorial memory task (on-line) 1 second stimulation and 14 seconds inter-train interval for 76 trains resulting in a total of 1520 pulses.
  Arms: High frequency Active control
Device: rTMS (low frequency active control ) — * Frequency: 1 Hz
  * Intensity: 110% of rMT
  * Location: Right superior frontal cortex of the dominant brain hemisphere
  * Duration: 6 minutes
  * Timing: Starting 1 minutes before and continuing during the memory task (Online)
  Arms: Low frequency Active control
Device: rTMS ( cTBS 30 Hz active control) — * Bilateral continuous theta burst stimulation (cTBS) 30 Hz:
  * Frequency: trains of 30 Hz (3 pulses) every 167 ms (frequency of 6 Hz, in the range of theta band)
  * Intensity: 100% of resting motor threshold (rMT)
  * Location: consecutively on right superior frontal cortex
  * Duration: 33.3 seconds for each side
  * Timing: Immediately before pictorial memory task (off-line)
  Arms: cTBS 30 Hz Active control
Device: rTMS (cTBS 30 Hz) — * Bilateral continuous theta burst stimulation (cTBS) 30 Hz:
  * Frequency: trains of 30 Hz (3 pulses) every 167 ms (frequency of 6 Hz, in the range of theta band)
  * Intensity: 100% of resting motor threshold (rMT)
  * Location: consecutively on left and right temporo-occipital cortex
  * Duration: 33.3 seconds for each side
  * Timing: Immediately before pictorial memory task (off-line)
  Arms: cTBS 30Hz

SUMMARY:
A pilot study, examining the effect of repeated transcranial magnetic brain stimulation (rTMS) on the formation of memories with negative valence. The investigators hypothesize that an effective rTMS protocol to reduce memory performance for adverse events can be found.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Generally healthy
* Normotensive (BP 90/60mmHg - 140/90mmHg)
* BMI: 19 - 30 kg/m2
* Age: 18 - 30 years
* Fluent German-speaking

Exclusion Criteria:

* Metal in the brain, skull or elsewhere in the body (e.g., splinters, fragments, clips, etc.)
* Implanted neurostimulator (e.g., DBS, epidural/subdural, VNS)
* Cardiac pacemaker or intracardiac lines
* Medication infusion device
* Nonremovable Piercings in the head area, pivot teeth (retainers are no exclusion criterion)
* Tattoos (head area) less than 3 months old or older than 20 years
* Condition after neurosurgery
* Hearing problems or tinnitus
* Not able to sit still due to tremor, tics, itching
* History of repeated syncope
* Head trauma diagnosed as concussion or associated with loss of consciousness
* diagnosis of epilepsy, or a convulsion or a seizure in the past of the participant or his/her close family
* TMS in the past showing problems
* Surgical procedures to spinal cord
* Spinal or ventricular derivations
* Alcohol or drug intake 48 hours before start of visits
* Regular intake of any medication or CNS-active medication 48h before visit
* rMT above the limits of rTMS device.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 105 (Actual)
Dates: Start 2023-06-06 (Actual); Primary Completion 2025-04-01 (Actual); Study Completion 2025-05-31 (Actual)

PRIMARY OUTCOMES:
memory recall performance | On average 1 hour after intervention
  The difference between valence specific (negative, positive, and neutral) memory performance as assessed by a standard picture recall episodic memory task.

SECONDARY OUTCOMES:
Working memory performance | On average 1 hour after intervention
  Working memory performance measured by n-back task

CONTACTS AND LOCATIONS:
Overall Officials: Dominique de Quervain, Prof. MD, Study Chair — University of Basel, Research Platform Molecular and Cognitive Neuroscience
Locations (1):
- University of Basel, Division of Cognitive Neuroscience, Basel, Canton of Basel-City, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
All IPD (de-identified) that underlie results in a publication will be shared upon reasonable request
Access Criteria: All IPD (de-identified) that underlie results in a publication will be shared upon reasonable request for scientific purposes. A reasonable request consists of a short description of the scientific purpose. Requests will be reviewed by the team of the principle investigator.